CLINICAL TRIAL: NCT03729089
Title: Predicting Fetal Outcome Using Third Trimester Modified Biophysical Profile Scan Compared to Standard of Care; an Open Label Randomized Controlled Trial at St. Francis Hospital Nsambya.
Brief Title: Third Trimester Modified Biophysical Profile Scan for Predicting Fetal Outcome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Andrew Odur (Other)
Collaborators: Uganda Martyrs University, St. Francis Hospital Nsambya, Jerusalem IHS and Andrew Abaasa (Study statistician) (Unknown)
Responsible Party: Sponsor-Investigator, Dr Andrew Odur, Resident (MMED) in Obstetrics and Gynecology, St. Francis Hospital Nsambya
Organization: St. Francis Hospital Nsambya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BPP-NSA-001
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Perinatal Death; Third Trimester Modified Biophysical Profile Scan
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: Eligible pregnant women at 34 to 40 weeks gestation will be randomized to interventional group (Biophysical profile scanning) or to a control group receiving the current standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Biophysical Profile scan (Experimental): Participants randomized to intervention group (modified biophysical profile scanning) will receive scans starting from 34 weeks at enrollment then every 3 weeks thereafter until 40 weeks of amenorrhea.
  Interventions: Other: Modified Biophysical Profile scan
- Current standard of care (No Intervention): The participants randomized to this control group will receive the current standard of care recommended by World Health Organization implemented by the attending Doctor. they may receive the modified biophysical profile scanning or not but at non specified time during their pregnancy.

INTERVENTIONS:
Other: Modified Biophysical Profile scan — Modified biophysical profile scan to be done in third trimester for eligible pregnant mothers
  Arms: Modified Biophysical Profile scan

SUMMARY:
Study topic:

Predicting fetal outcome using third trimester modified biophysical profile (BPP) scan compared with standard of care; a randomized clinical trial at St. Francis Hospital, Nsambya.

This is an open label randomized clinical trial comparing the third trimester modified biophysical profile done between 34 to 40 weeks with the current standard of care in reducing perinatal mortality at St. Francis Hospital, Nsambya

Objectives of the study:

Broad study objectives:

To evaluate the role of third trimester modified biophysical profile scan in predicting fetal outcome among pregnant mothers at St. Francis Hospital, Nsambya.

Specific study objectives:

* To determine the percentage decline in perinatal mortality following use of third trimester biophysical profile from 34 to 40 weeks at St. Francis Hospital, Nsambya.
* To determine if use of third trimester BPP scan improves prediction of perinatal outcome more than the current standard of care at St. Francis Hospital, Nsambya.
* To determine the fetal outcome of pregnancies done modified BPP and those who received current standard of care at St. Francis Hospital, Nsambya.

Hypothesis:

The hypothesis of the study is that performing third trimester modified biophysical profile scan between 34 and 40 weeks compared to standard of care is associated with a 16 percent reduction

DETAILED DESCRIPTION:
Randomization:

Eligible participants will be randomly allocated to one of the two study groups (modified biophysical profile scan arm or current standard of care arm) by an independent statistician who will not be involved in data analysis. The independent statistician will generate a randomization register consisting of the sequential study numbers but without the allocated study group. The register will be held at the enrollment clinic and patients who will be eligible for enrollment will be assigned the next available number on the register until the required sample size is reached. The principal investigator will identify a secure room from where opaque envelopes containing the different study arms will be kept. Participants will pick envelopes randomly from the pool of envelopes to obtain the study arm to which they automatically belong.

Blinding:

The study will be open label but only blinding the allocation at study entry.

Randomization concealment

No one including the independent statistician will know the study arm at the point of randomization. Because the intervention is not blinded, the rest of the study team including the principle investigator will get to know the study arm after the women have been randomized.

Sample size:

The use of fetal biophysical profile has been associated with 61 to 79 percent reduction in fetal mortality and morbidity. The incidence of perinatal death (Macerated still birth, Fresh stillbirth & Early neonatal death) in 2016 was 2% of the annual total deliveries, giving a perinatal mortality ratio of 20 per 1000 live birth at St. Francis Hospital Nsambya. The following assumptions will be made in the determination of the minimum sample size; the current standard of care of mothers attending antenatal care at Nsambya Hospital as defined by World health organization (WHO) in 2016 will detect up to 79% of fetal outcome, while performing modified biophysical profile scan proposed in this trial will increase this proportion to 95% at the 5% level of significance, and power of 80. Using a formula for comparing two proportions from Medical statistics book by Betty Kirkwood and Jonathan Sterne, 2003; The minimum sample size , Where this gives an increase in prediction of 16%. V= the Standard normal deviate at 95% Confidence (from Z-statistical tables, V=1.96), U =Standard Normal Deviate at 80% Power (power =1-β) ( from Z-statistical tables, u=0.84). Substituting, = 89.2 women. This gives approximately 90 women in each group and a total sample size of 180 women. Assuming a non-response proportion of 10%, the sample size will be increased by 10% to 198 women (99 in each group).

Data management and handling:

The study data will be entered using Microsoft (MS) access (MS-ACCESS, 2016) and will be double checked and validated before being uploaded into the database. The data entry screens will incorporate a number of range checks and logical skips as appropriate. Data stored in the database will be checked for missing or unusual values (range checks) and checked for consistency within participants. If any such problems are identified the problematic questionnaire will be returned to the clinic for checking and confirmation or correction, as appropriate. The amended version will be returned to the data entrant for correct entry into the database.

Statistical analysis plan:

Participant socio-demographics and other characteristics will be summarized using counts and percentages and by study group, for categorical variables and means and standard deviation for continuous variables. The analysis will be by intention to treat (ITT). I will calculate the mortality rate as the number of death divided by total time of follow up. The mortality will be further stratified by the study group (intervention vs standard of care). Rate ratio comparing the trial groups will be estimated by fitting a cox regression model. If there are any imbalance in the important participant characteristics at baseline, adjustment for these will be performed by fitting cox regression models. A similar analysis will be performed for the secondary outcomes.

Data quality control:

The study team will be trained on data collection and handling procedures. A pretest in form of completing the study questionnaire as well as a dry run will be done before the commencement of the actual data collection. To ensure proper data management, the data collectors will be trained in data management and will complete certification process of Good Clinical Practices (GCPs). Data collectors will be health workers who work in the Obstetrics department, they will not be directly involved in the management of mothers in Antenatal clinic or inpatient wards to avoid observation bias if he/she was among the people managing these patients. All interviews will be conducted in the language understood by the study participants.

Data monitoring committee:

There will be a data monitoring committee established to monitor the quality of data being collected. This three member committee will be selected from outside the study site. They will be people with experience in monitoring trial data. They will sit every 3 months or as requested by the institutional review board of St. Francis Hospital Nsambya.

Data protection and confidentiality:

The study questionnaires will not bear participant names but rather identification numbers. The study team will ensure the data is not accessible to anyone else by 1) keeping the paper questionnaires under lock and key 2) using passwords to secure the study database. The team will also ensure that the study data is used for only the purpose approved by the ethics committees.

Ethical considerations:

The study will seek ethical approvals from the Institutional Review Board (IRB) of Nsambya Hospital. The Hospital authority will also be requested for permission to have access to the pregnant women in the study clinic. Participants will be allowed to withdraw from the study whenever they so wish. All the data collected will be treated with utmost confidentiality.

STANDARD OPERATING PROCEDURE (SOP) FOR ENROLLMENT/SCREENING VISIT

1. The pregnant women are received, welcomed and briefed about the services by the midwife in the Antenatal clinic registration desk.
2. The midwife registering at the reception will identify pregnant women who are between 34 to 40 weeks gestation.
3. If one is attending for the first time but within the gestational age of interest, then the base line investigations will be done (Complete blood count, blood grouping, HIV, Urinalysis, Gestational diabetes mellitus screening, Syphilis test and Hepatitis B test).
4. For those who have been booked already, the study midwife will check the antenatal card and results of the above. If any is missing, a request would be written and sample taken.
5. Body weight and blood pressure will be measured at this point.
6. Immediately after receiving the antenatal card, the pregnant women will be directed to the waiting area from where routine antenatal health education and information about the study is given by one of the Antenatal clinic and study Midwives.
7. After providing information about the study, the study midwife will duly consent the mother and assign the randomization number sequentially from the register to those who volunteer to participate in the study.
8. The pregnant mother is accompanied by midwife to the study office (Room 9) from where the PI will request the mother to randomly pick an opaque envelope from the randomization pack to determine the study arm of this study participant.
9. The study arm will be known by the study team at this point and clearly documented in the patient's antenatal card.
10. The enrolled mothers will be examined by the study doctor or midwives and findings documented in the Antenatal card and Case report form (CRF).
11. The mothers in the modified Biophysical profile ARM will be required to undergo a modified biophysical profile scanning free of charge and the results of the scan documented in the CRF.
12. The mother will bring back the results of the scan and blood tests to the study doctor. The study doctor will document the above results on the CRF. He will give an appropriate follow up date and indicate the date for performing the next modified biophysical profile (mBPP) scan.
13. The registers and all other documents are taken to the research office at the end of the day by the Clinical Trial Midwife. All completed CRFs are scrutinized by the Trial PI and signed. If the Trial midwife detects errors in the CRFs, He or she will put a Note to the file accordingly as per the data management SOP.
14. The completed file folders will then be placed in the rack for not entered data. The entry into the data base will then be as per the data management SOP.

STANDARD OPERATING PROCEDURE FOR MISSED VISITS

1. The pre-enrollment and enrollment registers will have the scheduled appointments for each study participant.
2. Any study participant who fails to honor an appointment will be followed up with a phone call the next day to ascertain the reason why she did not turn up and encouraged to come. If she fails to turn up, a second phone call will be made and another appointment fixed.
3. A study participant who fails to honor her appointments and fails to respond to the above follow up would be considered as one lost to follow up.

STANDARD OPERATING PROCEDURE FOR TRACING MOTHERS WHO HAVE GONE PAST THEIR EXPECTED DATE OF DELIVERY (EDD) / DELIVERED ELSEWHERE

1. Each week, mothers who have not delivered at the study site are traced from the CRF/date of delivery list by the principle investigator.
2. The study participant is given a phone call and advised to visit the study site if not delivered to see the Doctors to assess her and plan for her delivery. If the person has already delivered from elsewhere, information regarding delivery is obtained and entered into the CRF.

STANDARD OPERATING PROCEDURE FOR UNSCHEDULED VISIT

1. Participants will be encouraged to come in every time they have a problem direct to Antenatal clinic Room 9 or labor ward in case it's after 5.00 pm where a doctor reviews her and the clinical trial coordinator is informed.
2. Participant will be seen by the Clinical Trial Investigator in the Antenatal Clinic on Monday- Friday from 8:00am-5:00pm.
3. After 5:00pm, during weekends, public holidays, Participant will report to the Labor ward and be seen by the Doctor on Duty and managed appropriately.

STANDARD OPERATING PROCEDURE FOR DOCUMENTING DELIVERY AND FETAL OUTCOME

1. Identification of study Participants who present in labor ward will be done by any of the labor ward midwives by asking for their antenatal card bearing the sticker and by asking whether the participant has been in the study. This process will be for both mothers in labor and those scheduled for Cesarean section.
2. The labor ward midwives will then inform one of the research midwives about the study participant. The research midwife will then verify the antenatal records and place an appropriate sticker on the patient file for easy identification. The study midwife will duly inform the Principle investigator.
3. For mothers who will undergo an elective or emergency cesarean section, the birth outcome will be documented from the post natal wards.
4. Immediately after delivery of the baby, the study midwife will document the birth outcome in the CRF which placed in a box file awaiting data cleaning and entry.
5. The above procedure will be followed for delivery during day, night and over the weekend.

STANDARD OPERATING PROCEDURE FOR DATA MANAGEMENT

1. The Case report form (CRF) will be assessed by the Clinical Trial Principle Investigator daily for accuracy, legibility and completeness.
2. The CRFs will then be filled, placed in the respective file folder and then placed in the rack for not entered data.
3. Only authorized study staffs (the Data Clerks, Principal Investigator, statisticians) are allowed to have access to the database.
4. Every afternoon, the Data Clerk will pick the CRFs from the box file of not entered data and then enter it into the database (Epi-data)
5. At the end of the day, all data will be saved and backed up on a flash disk or External Hard Drive.
6. After the CRFs have been entered into the database, they will be placed in the Box file for entered data for proper storage by one of the Data Clerks.

STANDARD OPERATING PROCEDURE FOR COMPLETING CASE REPORT FORM (CRF)

1. CFR must be filled with a ball-point-black ink.
2. Capital letters must be used in all entries of the CRF. The dates that are not known will be represented with value 11/11/1111.
3. The Principle investigator and the Trial Coordinator will write Not applicable on all different CRF for non obtainable information whether numerical or non numerical.
4. Corrections on CRF will be done by the person who has filled in that CRF.
5. Corrections will be done by crossing out the wrong entry with a single line, then writing the correct entry alongside/above/under the wrong entry.
6. After correction, a date will be placed alongside the correction as well as the initials of the Research staff.
7. A note to file will be placed on that page of the CRFs to explain the correction by the Research staff and confirmed by the Principal investigator

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton pregnancy
* Gestational age between 34 to 40 weeks based on reliable date of onset of last normal menstrual period or earliest dating by ultrasonography.
* Willing to be followed up

Exclusion Criteria:

* Mother with diagnosed fetal malformations
* High-risk pregnancies (Hypertensive disorders of pregnancy, Diabetes mellitus, multiple pregnancies, Sickle cell disease, Heart disease).
* Inability to consent (e.g. psychiatric conditions or very ill requiring hospitalization).
* Intrauterine fetal death in the current pregnancy
* Presently ill with a medical condition requiring admission to hospital

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Perinatal death | At delivery of the newborn
  Reduction in the proportion of perinatal death will be measured for the two arms of the study to ascertain whether modified biophysical profile can predict perinatal mortality. Perinatal mortality will be measured as death of the new born within the first 7 days of life. The gestational age considered is after 28 weeks of amenorrhea consistent with the health system capacity of the host country and the study hospital

SECONDARY OUTCOMES:
APGAR score | at birth
  The APGAR score is a clinical score used to assess well being of all newborns. The clinical features of newborn colour, Respiration, Heart rate, muscle tone and reflex stability depends on the aetiology, intensity and duration of oxygen lack, plasma carbondioxide excess and subsequent acidosis. The score will be taken at 1 minute and at 5 minutes after birth and documented in the case report form. Minimum score is 0/10 while the maximum is 10/10. A score of less than 3/10 at 5 minutes indicates severe birth asphyxia; a score of 4/10 to 6/10 signifies moderate asphyxia and 7/10 to 10/10 is a normal new born. The higher the score, the better the neonatal outcome.
Neonatal intensive care unit (NICU) admission | Immediately after birth
  The neonatal intensive care (NICU) admission of the newborn will be documented as yes or no at birth. This will be assessed by documenting the post delivery decision of the attending health worker on whether the baby needs NICU admission or not
Cesarean section due to fetal condition | At delivery
  Cesarean section (C/S) performed for fetal conditions will be assessed by the study team by looking out for the indication of C/S and document if it was done due to fetal conditions like non reassuring fetal status, meconium stained liquor, severe oligohydramnios, cord accidents and abnormal fetal heart pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Odur, MBChB, DPPM, Principal Investigator — St. Francis Hospital Nsambya; Romano Byaruhanga, MMed, PhD, Study Chair — St. Francis Hospital Nsambya; Rita Nassanga, MMed, Study Chair — St. Francis Hospital Nsambya; Gilbert Tumwine, MMed, MPH, Study Chair — St. Francis Hospital Nsambya
Locations (1):
- St. Francis Hospital Nsambya, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Only data necessary for publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after publication
Access Criteria: Data will be accessed for now on request from the Principle investigator and shared through email